CLINICAL TRIAL: NCT04823169
Title: Painful and Barometric Dynamic Monitoring in the Aftermath of Foot Surgery Using the Distal Metatarsal Mini-invasive Osteotomy (DMMO) Method.
Acronym: BAROC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHM-2020/S11/09
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Distal Metatarsal Mini-invasive Osteotomy (DMMO)
Keywords: Distal Metatarsal Mini-invasive Osteotomy; DMMO; Podobarometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- podobarometry (Experimental): podobarometric measures at day7 and day 30
  Interventions: Other: podobarometry

INTERVENTIONS:
Other: podobarometry — podobarometric measures on day 7 and day 30

SUMMARY:
The definitive treatment of disabling metatarsalgia requires surgery. In recent years, a percutaneous technique has been developed, the "Distal Metatarsal Mini-invasive Osteotomy" (DMMO). It consists of performing extra-articular osteotomies that are not osteosynthesized and maintained during the time of bone consolidation by a dressing and specific offloading footwear.The patient is encouraged to resume walking immediately after the procedure, as full plantar support is an integral part of the surgical concept. The goal is to actively modify the distribution of all metatarsal supports by the pressure exerted on the ground during walking and by tendon tensions, in order to reduce forefoot deformities.

DMMO offers many advantages over traditional techniques, but it remains a painful forefoot surgery in the short term despite the systematic use of analgesics and the wearing of a dedicated therapeutic shoe.

The study will seek to identify the predictive character of podobarometric parameters at walking (D+7 and D+30 post-op), between patients who will require a palliative solution versus those who will not (D+90)

ELIGIBILITY:
Inclusion Criteria:

* Adult person
* Affiliated or beneficiary of a statutory social insurance scheme
* Free ans informed consent
* Following foot surgery like DMMO only or DMMO and hallux valgus

Exclusion Criteria:

* Minor or legally protect adult
* Amputation disturbing the natural course of the step
* Osteoarticular diseases/sequelae affecting walking and/or balance
* Neuromuscular diseases/sequelae affecting walking and/or balance
* Vestibular disorders affecting balance
* Patients requiring a walking aid (e.g., walker)
* Pregnant woman
* Patient with dementia who are unable to follow verbal instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-09-22 (Estimated); Study Completion 2023-09-22 (Estimated)

PRIMARY OUTCOMES:
podobarographic parameters (plantar pressures) predictive of the need for a palliative foot orthosis | 90 days after surgery
  Plantar pressures were measured by podobarometric Platform (FREEMED Platform)

SECONDARY OUTCOMES:
Compare daily walk pain kinetics over one month postoperatively in patients requesting palliative solutions at 3 months (requesters) versus those not requesting them (non-requesters) | 90 days after surgery
  Daily walk pain was measured by questionnaire (Google form) completed by patient every day during 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France